CLINICAL TRIAL: NCT00525798
Title: A Randomized, Double-Blind, Multi-Center, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Oral Salmon Calcitonin in the Treatment of Osteoporosis in Postmenopausal Women Taking Calcium and Vitamin D
Brief Title: A Study to Evaluate Oral Salmon Calcitonin in the Treatment of Osteoporosis in Postmenopausal Women Taking Calcium and Vitamin D
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nordic Bioscience A/S (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMC021A2303
Record Dates: First submitted 2007-09-05; First posted 2007-09-06 (Estimated); Results first posted 2012-10-18 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: Osteoporosis
Keywords: Osteoporosis, oral salmon calcitonin, treatment, efficacy, tolerability
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): SMC021 - Oral Calcitonin
  Interventions: Drug: SMC021 Oral calcitonin
- SMC021- Placebo (Placebo Comparator): SMC021 - placebo
  Interventions: Drug: SMC021 Placebo

INTERVENTIONS:
Drug: SMC021 Oral calcitonin — 0.8mg SMC021 - oral calcitonin, once daily
  Arms: 1
Drug: SMC021 Placebo — SMC021 - Placebo, once daily
  Arms: SMC021- Placebo

SUMMARY:
The purpose of this Phase III study is to evaluate the efficacy and safety of oral salmon calcitonin in the treatment of patients with osteoporosis

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with osteoporosis, ambulatory, in general good health, not receiving medication that affects bone metabolism, and free from any underlying condition, other than osteoporosis, that may result in abnormal bone metabolism.

Exclusion Criteria:

* BMD T-score below -4.0 (based on absolute values g/cm2 as given in the protocol) at one or more of the measured sites
* More than 2 prevalent vertebral fractures (Genant et al, 15).
* If BMD is lower than -2.5 T-score at one or more of the measured sites, the participants will be excluded from the study, if they have a severe vertebral fracture (Genant et al, 15).
* Evidence of any clinical osteoporotic fracture and/or if they have a history of a clinical osteoporotic fracture (excluding wrist fractures)
* BMD T-score > -1.5 in all of the following regions: Lumbar spine, femoral neck or total hip.

Other protocol defined inclusion/exclusion criteria may apply

Ages: 55 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4665 (Actual)
Dates: Start 2007-03; Primary Completion 2011-08 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bente J Riis, M.D., Study Chair — Nordic Bioscience A/S
Locations (16):
- United States (3):
  - United Osteporosis Centers, Gainesville, Georgia
  - Michigan Bone & Mineral Clinic PC,, Detroit, Michigan
  - Oregon Osteoporosis Center, Portland, Oregon
- CCBR Brazil, Rio de Janeiro, Brazil
- CCBR China, Beijing, China
- CCBR Czech, Pardubice, Czechia
- Denmark (3):
  - CCBR Aalborg, Aalborg
  - CCBR Ballerup, Ballerup Municipality
  - CCBR Vejle, Vejle
- CCBR Estonia, Tallinn, Estonia
- Hopital Edouard Herriot, Lyon, France
- CCBR Hong Kong, Hong Kong, Hong Kong
- Department of Internal Medicine, University of Florence, Florence, Italy
- CCBR Lithuania, Vilnius, Lithuania
- CCBR Poland, Warsaw, Poland
- CCBR Romania, Bucharest, Romania

REFERENCES:
- [Derived] Henriksen K, Bay-Jensen AC, Christiansen C, Karsdal MA. Oral salmon calcitonin--pharmacology in osteoporosis. Expert Opin Biol Ther. 2010 Nov;10(11):1617-29. doi: 10.1517/14712598.2010.526104. Epub 2010 Oct 11. PMID 20932224

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at 16 centers in 12 countries:
  3 centers in the US and 3 centers in Denmark.
  1 center in Brazil, Estonia, Czech Republic, Poland, Lithuania, Romania, Italy, France, Hong Kong, and China.
  First patient randomized: 26 Feb 2007 Last patient visit: 30 Jul 2011
Groups:
- SMC021: 1 tablet of 0,80 mg SMC021 daily
- Placebo: 1 tablet of placebo daily
Period: Overall Study
Arm/Group | SMC021 | Placebo
Started | 2334 | 2331
Completed | 1578 | 1732
Not Completed | 756 | 599

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SMC021 | Placebo | Total
Number analyzed (Participants) | 2334 | 2331 | 4665
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 912 | 860 | 1772
  >=65 years | 1422 | 1471 | 2893
Age Continuous [Mean (Standard Deviation); unit: years] | 66.5 (6.12) | 67.0 (6.16) | 66.8 (6.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2334 | 2331 | 4665
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 31 | 30 | 61
  France | 2 | 2 | 4
  Hong Kong | 74 | 73 | 147
  Czech Republic | 230 | 232 | 462
  Estonia | 167 | 166 | 333
  Brazil | 492 | 492 | 984
  Poland | 176 | 176 | 352
  Lithuania | 149 | 150 | 299
  Romania | 172 | 171 | 343
  Denmark | 599 | 598 | 1197
  Italy | 18 | 17 | 35
  China | 224 | 224 | 448

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With New Vertebral Fractures
Description: The primary variable was the occurrence or not of a new vertebral fracture during the 3 year observation period. New vertebral fractures were identified from an assessment of x-ray of the lateral spine through time (at baseline and at yearly intervals thereafter).
  The outcome is the number of new vertebral fractures from baseline to 36 months.
Time Frame: From baseline to month 36
Population: all patients randomized who received at least one dose of study drug, with the addition of evaluable baseline spine X-ray and at least one follow-up for calculation of vertebral fractures.
Measure: Number; unit: Participants
Arm/Group | SMC021 | Placebo
Number analyzed (Participants) | 2064 | 2125
Participants | 94 | 99

2. Secondary Outcome: Number of Patients With Non-vertebral Fractures
Description: The secondary outcome was the occurrence or not of a non-vertebral fracture during the 3 year observation period. Non-vertebral fractures of interest were: hip fractures, forearm fractures, humurus fractures, rib fractures and clavicular fractures.
  Any new non-vertebral fractures while on-study were recorded. A copy of radiographs confirming the fracture, as well as a copy of the radiologist's report was to be obtained. A copy of the emergency room discharge letter or a hospital discharge letter was also obtained.
Time Frame: From baseline to month 36
Population: all randomized patients
Measure: Number; unit: Participants
Arm/Group | SMC021 | Placebo
Number analyzed (Participants) | 2334 | 2331
Participants | 75 | 82

ADVERSE EVENTS:
Time Frame: From baseline to 36 month
Arm/Group | SMC021 | Placebo
Serious Adverse Events (participants affected / at risk) | 340/2334 | 378/2331
Other Adverse Events (participants affected / at risk) | 2152/2334 | 2141/2331
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SMC021 (N=2334) | Placebo (N=2331)
Anemia (Blood and lymphatic system disorders) | 0 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 10 | 8
Acute myocardial infarction (Cardiac disorders) | 6 | 3
Coronary artery disease (Cardiac disorders) | 5 | 5
Angina pectoris (Cardiac disorders) | 5 | 4
Myocardial ischaemia (Cardiac disorders) | 4 | 3
Angina unstable (Cardiac disorders) | 3 | 6
Myocardial infarction (Cardiac disorders) | 3 | 4
Arrhytmia (Cardiac disorders) | 3 | 1
Cardiac failure (Cardiac disorders) | 3 | 1
Cardiac failure congestive (Cardiac disorders) | 3 | 0
Atrial flutter (Cardiac disorders) | 2 | 2
Arteriosclerosis coronary artery (Cardiac disorders) | 2 | 0
Aortic valve stenosis (Cardiac disorders) | 1 | 1
Sick sinus syndrome (Cardiac disorders) | 1 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Aortic valve disease (Cardiac disorders) | 0 | 1
Bundle branch block left (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Coronary artery dilatation (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Coronary artery thrombosis (Cardiac disorders) | 0 | 1
Hypertrophic cardiomyopathy (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Ventricular dysfunction (Cardiac disorders) | 0 | 1
Ventricular failure (Cardiac disorders) | 0 | 1
Hereditary haemorrhagic telangiectasia (Congenital, familial and genetic disorders) | 1 | 0
Abdominal wall anomaly (Congenital, familial and genetic disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 3
Deafness (Ear and labyrinth disorders) | 1 | 0
Meniere´s disease (Ear and labyrinth disorders) | 1 | 0
Otosclerosis (Ear and labyrinth disorders) | 1 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Vestibular ataxia (Ear and labyrinth disorders) | 0 | 1
Goitre (Endocrine disorders) | 2 | 2
Hypothyroidism (Endocrine disorders) | 1 | 0
Thyroid disorder (Endocrine disorders) | 1 | 0
Hypothyroidic goitre (Endocrine disorders) | 0 | 1
Cataract (Eye disorders) | 6 | 3
Glaucoma (Eye disorders) | 2 | 1
Retinal detachment (Eye disorders) | 1 | 1
Macular degeneration (Eye disorders) | 1 | 0
Maculopathy (Eye disorders) | 1 | 0
Scleritis (Eye disorders) | 1 | 0
Eye disorder (Eye disorders) | 0 | 2
Angle closure glaucoma (Eye disorders) | 0 | 1
Optic atrophy (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Inguinal hernia (Gastrointestinal disorders) | 3 | 0
Abdominal hernia (Gastrointestinal disorders) | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 2
Ileus (Gastrointestinal disorders) | 2 | 2
Haemorrhoids (Gastrointestinal disorders) | 2 | 1
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Colonic polyp (Gastrointestinal disorders) | 1 | 4
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2
Colitis (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 1
Femoral hernia (Gastrointestinal disorders) | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1
Coeliac disease (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Enterocele (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Lumbar hernia (Gastrointestinal disorders) | 1 | 0
Mechanical ileus (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 2
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Intussusception (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Rectal polyp (Gastrointestinal disorders) | 0 | 1
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 3 | 8
Death (General disorders) | 3 | 2
Pyrexia (General disorders) | 2 | 0
Adverse drug reaction (General disorders) | 1 | 0
Device occlusion (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Thrombosis in device (General disorders) | 1 | 0
Chest discomfort (General disorders) | 0 | 2
Accidental death (General disorders) | 0 | 1
Sudden cardiac death (General disorders) | 0 | 1
Ulcer (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 19 | 9
Cholecystitis acute (Hepatobiliary disorders) | 2 | 2
Cholecystitis chronic (Hepatobiliary disorders) | 2 | 0
Gallbladder polyp (Hepatobiliary disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 2
Biliary colic (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Pneumonia (Infections and infestations) | 12 | 11
Diverticulitis (Infections and infestations) | 3 | 3
Appendicitis (Infections and infestations) | 3 | 1
Urinary tract infection (Infections and infestations) | 2 | 2
Bronchitis (Infections and infestations) | 1 | 3
Gastroenteritis (Infections and infestations) | 1 | 2
Pyelonephritis (Infections and infestations) | 1 | 2
Septic shock (Infections and infestations) | 1 | 1
Urosepsis (Infections and infestations) | 1 | 1
Bacterial infection (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Encephalitis viral (Infections and infestations) | 1 | 0
Gallbladder empyema (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 1 | 0
Hepatitis C (Infections and infestations) | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 1 | 0
Perineal infection (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 2
Herpes zoster (Infections and infestations) | 0 | 2
Bronchopneumonia (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Neurological infection (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 0 | 1
Pelvic inflammatory disease (Infections and infestations) | 0 | 1
Pyometra (Infections and infestations) | 0 | 1
Salmonellosis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Vaginal infection (Infections and infestations) | 0 | 1
Viral pericarditis (Infections and infestations) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 8 | 8
Femoral neck fracture (Injury, poisoning and procedural complications) | 5 | 3
Humurus fracture (Injury, poisoning and procedural complications) | 4 | 4
Femur fracture (Injury, poisoning and procedural complications) | 3 | 9
Concussion (Injury, poisoning and procedural complications) | 3 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 2 | 3
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 2
Radius fracture (Injury, poisoning and procedural complications) | 2 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 4
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0
Avulsion fracture (Injury, poisoning and procedural complications) | 1 | 0
Burns secound degree (Injury, poisoning and procedural complications) | 1 | 0
Burns third degree (Injury, poisoning and procedural complications) | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 | 0
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0
Perineal laceration (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 3
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 3
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 2
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 2
Rib fracture (Injury, poisoning and procedural complications) | 0 | 2
Wound (Injury, poisoning and procedural complications) | 0 | 2
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Postoperative hernia (Injury, poisoning and procedural complications) | 0 | 1
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 0 | 1
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 2 | 1
International normalised ratio increased (Investigations) | 1 | 0
Arteriogram coronary (Investigations) | 0 | 1
Arthroscopy (Investigations) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 19 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 3 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 2 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 | 0
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 2 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 | 12
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Adult T-cell lymphoma/leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometríal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lipoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nasal cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamos cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adrenocortical carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carcinoid tumour of the stomach (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervix carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrooesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mucoepidermoid carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Spinal haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 10 | 8
Ischaemic stroke (Nervous system disorders) | 5 | 5
Syncope (Nervous system disorders) | 3 | 4
Transient ischaemic attack (Nervous system disorders) | 2 | 9
Headache (Nervous system disorders) | 1 | 3
Reversible ischaemic neurological deficit (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 1
Loss of consciousness (Nervous system disorders) | 1 | 1
Brain stem infarction (Nervous system disorders) | 1 | 0
Brain stem thrombosis (Nervous system disorders) | 1 | 0
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0
Diabetic neuropathy (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Trigeminal neuralgia (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 4
Cerebral thrombosis (Nervous system disorders) | 0 | 3
Amnesia (Nervous system disorders) | 0 | 2
Epilepsy (Nervous system disorders) | 0 | 2
Haemorrhagic stroke (Nervous system disorders) | 0 | 2
Hypertensive encephalopathy (Nervous system disorders) | 0 | 2
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebrovascular disorder (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
IIIrd nerve paralysis (Nervous system disorders) | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 0 | 1
Paralysis (Nervous system disorders) | 0 | 1
Parkinsonism (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 0 | 1
Vascular dementia (Nervous system disorders) | 0 | 1
Vertebral artery stenosis (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 2 | 2
Cystitis noninfective (Renal and urinary disorders) | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 1
Renal cyst (Renal and urinary disorders) | 1 | 1
Bladder prolapse (Renal and urinary disorders) | 1 | 0
Bladder disorder (Renal and urinary disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Urethral caruncle (Renal and urinary disorders) | 0 | 1
Urethral polyp (Renal and urinary disorders) | 0 | 1
Urinary bladder polyp (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Cystocele (Reproductive system and breast disorders) | 2 | 4
Uterine polyp (Reproductive system and breast disorders) | 2 | 3
Rectocele (Reproductive system and breast disorders) | 2 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 | 1
Uterine prolapse (Reproductive system and breast disorders) | 1 | 5
Vaginal prolapse (Reproductive system and breast disorders) | 1 | 2
Endometrial disorder (Reproductive system and breast disorders) | 1 | 0
Hydrometra (Reproductive system and breast disorders) | 1 | 0
Breast enlargement (Reproductive system and breast disorders) | 0 | 1
Genital disorder female (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Breast prothesis user (Social circumstances) | 0 | 1
Joint prothesis user (Social circumstances) | 0 | 1
Knee arthroplasty (Surgical and medical procedures) | 3 | 3
Hip arthroplasty (Surgical and medical procedures) | 3 | 2
Varicose vein operation (Surgical and medical procedures) | 3 | 0
Appendicectomy (Surgical and medical procedures) | 2 | 2
Mastectomy (Surgical and medical procedures) | 1 | 1
Wrist surgery (Surgical and medical procedures) | 1 | 1
Bone operation (Surgical and medical procedures) | 1 | 0
Oophorectomy bilateral (Surgical and medical procedures) | 1 | 0
Vaginaplasty (Surgical and medical procedures) | 1 | 0
Vascular graft (Surgical and medical procedures) | 1 | 0
Cataract operation (Surgical and medical procedures) | 0 | 7
Aortic bypass (Surgical and medical procedures) | 0 | 1
Breast prothesis removal (Surgical and medical procedures) | 0 | 1
Cardiac pacemaker battery replacement (Surgical and medical procedures) | 0 | 1
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 | 1
Cardiac pacemaker replacement (Surgical and medical procedures) | 0 | 1
Cholecystectomy (Surgical and medical procedures) | 0 | 1
Fracture reduction (Surgical and medical procedures) | 0 | 1
Gallbladder operation (Surgical and medical procedures) | 0 | 1
Genitourinary operation (Surgical and medical procedures) | 0 | 1
Haemorrhoid operation (Surgical and medical procedures) | 0 | 1
Hospitalisation (Surgical and medical procedures) | 0 | 1
Osteosynthesis (Surgical and medical procedures) | 0 | 1
Percutaneous coronary intervention (Surgical and medical procedures) | 0 | 1
Radical hysterectomy (Surgical and medical procedures) | 0 | 1
Hypertension (Vascular disorders) | 5 | 4
Varicose vein (Vascular disorders) | 3 | 2
Arteriosclerosis (Vascular disorders) | 2 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 1
Femoral arterial stenosis (Vascular disorders) | 2 | 0
Aneurysm (Vascular disorders) | 1 | 0
Arterial occlusive disease (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0
Temporal arteritis (Vascular disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 2
Aortic occlusion (Vascular disorders) | 0 | 1
Arteriosclerosis obliterans (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
Vasculitis (Vascular disorders) | 0 | 1
Shoulder operation (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SMC021 (N=2334) | Placebo (N=2331)
Nausea (Gastrointestinal disorders) | 357 | 117
Back Pain (Musculoskeletal and connective tissue disorders) | 311 | 339
Arthralgia (Musculoskeletal and connective tissue disorders) | 284 | 320
Hot flush (Vascular disorders) | 263 | 41
Nasopharyngitis (Infections and infestations) | 262 | 269
Hypertension (Vascular disorders) | 238 | 267
Dyspepsia (Gastrointestinal disorders) | 228 | 129
Constipation (Gastrointestinal disorders) | 165 | 172
Diarrhea (Gastrointestinal disorders) | 157 | 120
Abdominal pain upper (Gastrointestinal disorders) | 153 | 107
Hypercholesterolemia (Metabolism and nutrition disorders) | 137 | 149
Pain in extremity (Musculoskeletal and connective tissue disorders) | 136 | 186
Influenza (Infections and infestations) | 133 | 160
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 129 | 142
Erythema (Skin and subcutaneous tissue disorders) | 123 | 14
Dizziness (Nervous system disorders) | 120 | 105
Hypertriglyceridemia (Metabolism and nutrition disorders) | 118 | 120
Abdominal discomfort (Gastrointestinal disorders) | 114 | 57
Bronchitis (Infections and infestations) | 104 | 127
Pneumonia (Infections and infestations) | 102 | 108
Cystitis (Infections and infestations) | 100 | 96
Urinary tract infection (Infections and infestations) | 88 | 95
Cough (Respiratory, thoracic and mediastinal disorders) | 79 | 88
Headache (Nervous system disorders) | 72 | 80
Vomiting (General disorders) | 72 | 46
Anemia (Blood and lymphatic system disorders) | 69 | 77
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 66 | 82
Gastritis (Gastrointestinal disorders) | 64 | 57
Cataract (Eye disorders) | 63 | 84
Depression (Psychiatric disorders) | 62 | 58
Vertigo (Ear and labyrinth disorders) | 60 | 63
Contusion (Injury, poisoning and procedural complications) | 55 | 54
Viral infection (Infections and infestations) | 54 | 70
Abdominal distension (Gastrointestinal disorders) | 54 | 44
Hypocalcemia (Metabolism and nutrition disorders) | 53 | 33
Muscle spasms (Musculoskeletal and connective tissue disorders) | 47 | 42
Sinusitis (Infections and infestations) | 46 | 52
Insomnia (Psychiatric disorders) | 45 | 60
Edema peripheral (General disorders) | 44 | 63
Wrist fracture (Injury, poisoning and procedural complications) | 42 | 47
Chest pain (General disorders) | 37 | 69
Upper respiratory tract infection (Infections and infestations) | 35 | 48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days